CLINICAL TRIAL: NCT06547541
Title: Exercise Training During Hospitalization in Patients With Type 2 Diabetes - A Phase 1 Trial
Brief Title: Pilot - Resistance Exercise for Inpatient Treatment in T2D
Acronym: P-REFIT-T2D
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Too low recruitment.
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: TrygFonden, Denmark (Industry)
Responsible Party: Principal Investigator, Julie Abildgaard, Senior Researcher, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-24002354; PREFIT-T2D (Other: Centre for Physical Activity Research)
Record Dates: First submitted 2024-07-28; First posted 2024-08-09 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 2; Prediabetes or Diabetes; Prediabetes
Keywords: Exercise; Glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Diabetes Mellitus; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): The exercise intervention is a four-week intervention and will consist of body weight strength training. All training sessions during hospitalization will be supervised and will be performed individually for 30 min/day. If the patient is discharged within the four-week training period, the training will continue from home and will be online-based with a live video connection to an instructor. The training program will be the same. The intervention group will ideally exercise post-prandially (within 60 min following the meal) following either breakfast or lunch. Exercise intensity will be monitored throughout the training (with a heart rate monitor) and patients will estimate the rigorousness of the training using the rate of perceived exertion (RPE)-scale. If possible, the goal is for the patients to reach a minimum of 5, corresponding to moderate intensity, but preferably 7+ on the 0-10 RPE scale in each set. The aim is to complete the training sessions five out of seven days/week.
  Interventions: Behavioral: Exercise
- Control (No Intervention): The Control group will be placed in a chair for 30 minutes, within 60 minutes following either breakfast or lunch daily during admission, depending on other workflows in the ward. This corresponds to the time spent on exercise by the intervention group. The control group will also be in daily contact with the instructor following discharge and will be asked the same daily questions and will be seated in a chair for 30 minutes as during hospitalization.

INTERVENTIONS:
Behavioral: Exercise — A body weight based resistance training.
  Arms: Exercise

SUMMARY:
Type 2 Diabetes (T2D) is associated with prolonged hospitalization and an increased risk of readmission. Moreover, sedentary behavior and poor glycemic control may contribute to disease severity and mortality. The inactivity during hospitalization is particularly concerning in T2D patients, due to the negative effect on glucose metabolism and secondary loss of skeletal muscle mass, which can further disrupt glucose regulation. However, there are no exercise guidelines for hospitalized T2D patients. To address this gap, a feasibility study will be conducted examining the effectiveness of incorporating resistance training into hospital care for T2D patients. For the feasibility study, 24 patients with T2D or prediabetes will be recruited from the Department of Infectious Diseases at Rigshospitalet and Hvidovre Hospital and randomized to 4 weeks of resistance training for 30 minutes per day or standard treatment. If the participants are discharged they will be offered online-training sessions. During the hospitalization a continuous glucose monitor will be applied and an accelerometer during the full intervention. At baseline, discharge and at follow-up, extensive testing will be performed.

DETAILED DESCRIPTION:
Patients will be invited to participate, preferably within the first 24 hours of admission, and randomized to either resistance-based bodyweight exercise or a control group. In total, 24 patients will be recruited, and distributed between the groups stratified for biological sex. At baseline, participants will have their medical history, social anamnesis, height, and weight assessed. At baseline a continuous glucose monitor will and accelerometer will be applied, to be worn until discharge and end of the intervention, respectively. Furthermore at baseline a multitude of questionnaires will be performed: International Physical Activity Questionnaire (IPAQ), Strength, Assistance in walking, Rise from a chair, Climb stairs, and Falls (SARC-F), Brief Illness Perception Questionnaire (BIPQ), 5-level EQ-5D version (EQ-5D-5L), WHO-5 Well-Being Index (WHO-5).

Intervention session A body-weight based resistance exercise program will be performed based on a booklet "Syg men sund og aktiv" Sick but healthy and active for 30 minutes per day. Described in more detail below.

Control session The control group will be placed in a seated position for 30 minutes corresponding to the time the intervention group is active.

Assessments before and after intervention/control sessions Before the sessions the EQ-5D-5L, the WHO-5 modified to a daily version, and an acute assessment of malaise, tiredness, nausea, dizziness, pain and breathlessness will be performed using numerical rating scales (NRS). After the session the NRS will be performed again.

Follow-up visit Two days after completion of the intervention, the participants will be invited for a follow-up visit at the Centre for Physical Activity Research, Rigshospitalet. This visit includes a qualitative interview, assessment of body composition, assessment of physical capabilities, ultrasound of the thigh, and blood samples. In case the patient is unable to attend the follow-up visit at the center, the daily operating manager will visit the patient at home. In this case, Ultrasound and muscle biopsy will not be performed. If the patient lives more than one hour away by car, the assessment will be performed online and will not include ultrasound, body composition and blood tests.

ELIGIBILITY:
Inclusion Criteria:

* T2D or prediabetes defined as at least one of the following

  * ICD-10 diagnosis of T2D (DE11.x)
  * HbA1c > 48 at time of admission
  * Use of type 2 antidiabetic medicine (excluding SGLT2 inhibitors)
  * HbA1c ≥ 42 within 3 months of admission (prediabetes) (from 18 of September, 2024)
* Hospitalized with an infection
* Expected residual hospitalization time of at least three days
* At least 18 years of age
* Able to perform exercises in the booklet "Syg men sun dog aktiv"

Exclusion Criteria:

* Admitted to the hospital more than 5 days ago
* Unable to give written consent to participate
* Terminal illness
* Unstable or new onset angina
* Ventricular arrhythmia
* Aortic stenosis
* Sternotomy in conjunction with the current hospitalization
* Blood pressure greater than 180/120 mmHg
* Kidney failure requiring dialysis
* Unable to follow the 3-stage command of the Mini-Mental State Examination
* Known allergy or contact dermatitis to tape, and CGMs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2024-08-12 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Feasibility of exercise in hospitalized patients with type 2 diabetes | Baseline to follow-up visit (4 weeks).
  • Recruitment: Include 24 patients in five months. Failure to achieve this goal will indicate challenges in the recruitment process. The recruitment will be continuously evaluated.
  o Failure to recruit 5 participants within the 1st month of recruitment will lead to patients with prediabetes (HbA1c ≥ 42 mmol/mol) being eligible for inclusion. This criterion will be assessed monthly and if the projected recruitment of 4-5 patients/month is not met, the inclusion criteria will be expanded to include prediabetes. If so, an amendment will be submitted to change the title of the project to include prediabetes. An intermediate state of diabetes also has a higher frequency of critical outcomes during hospitalization, and is inversely related to skeletal muscle mass.
Glycemic variability | Baseline until discharge, with a maximum of 4 weeks post-inclusion.
  Coefficient of variance (%CV) during hospitalization evaluated using a continuous glucose monitor.
  Defined as the oscillations in blood glucose occurring throughout the day. High glycemic variability is associated with an increased risk of cardiovascular events, mortality, and impaired quality of life. Glycemic variability adds considerable nuance to blood glucose control and allows for short-term assessments compared to glycated hemoglobin. If the participant is not discharged after 4 weeks the data collection will stop.

SECONDARY OUTCOMES:
Short physical performance battery | Baseline to follow-up visit (4 weeks).
  The Short Physical performance battery (SPPB) will be assessed at baseline, discharge and 30-day follow-up. The SPPB consists of a combined score of a balance test (with the feet together, in a semitandem and tandem position), a walking test measuring the average speed over a three-meter distance, and a chair raise test that evaluates the time it takes for the participant to stand up and sit down five times.
Sit-down stand-up test | Baseline to follow-up visit (4 weeks).
  A sit down stand-up test will be performed at baseline, discharge and 30-day follow-up to assess the number of times the participant can stand up and sit down from a chair within 60 seconds.
Grip strength | Baseline to follow-up visit (4 weeks).
  Grip strength will be assessed at baseline, discharge and 30-day follow-up. Measurements will be taken three times per hand, with the participant in a seated position. The upper arm will be parallel to the torso, the elbow flexed at 90 degrees, and the wrist in a neutral position.
Duration of hospitalization | Baseline until discharge, with a maximum of 1 year post intervention.
  Number of days in hospital, from baseline until a maximum of 1 year post intervention.
Insulin use during hospitalization | Baseline until discharge, with a maximum of 4 weeks post-inclusion.
  Number of daily units during hospitalization, from baseline until a maximum of 4 weeks.
Mean glucose levels | Baseline until discharge, with a maximum of 4 weeks post-inclusion.
  Mean glucose levels during hospitalization assessed using a continuous glucose monitor.
  If the participant is not discharged after 4 weeks the data collection will stop.
Time in hyperglycemia | Baseline until discharge, with a maximum of 4 weeks post-inclusion.
  Time in hyperglycemia (blood glucose > 10 mmol/l) during hospitalization assessed using a continuous glucose monitor.
  If the participant is not discharged after 4 weeks the data collection will stop.
Time in hypoglycemia | Baseline until discharge, with a maximum of 4 weeks post-inclusion.
  Time in hypoglycemia (blood glucose < 4 mmol/l) during hospitalization assessed using a continuous glucose monitor.
  If the participant is not discharged after 4 weeks the data collection will stop.
Time in normal glucose range | Baseline until discharge, with a maximum of 4 weeks post-inclusion.
  Time in normal range (6-10 mmol/l in accordance with Danish guidelines), during hospitalization assessed using a continuous glucose monitor.
  If the participant is not discharged after 4 weeks the data collection will stop.
Mean amplitude of glucose excursions | Baseline until discharge, with a maximum of 4 weeks post-inclusion.
  Mean amplitude of glucose excursions from peaks to nadirs that are > 1 SD of mean glucose, assessed during hospitalization assessed using a continuous glucose monitor. If the participant is not discharged after 4 weeks the data collection will stop.
Cognitive function | Baseline to follow-up visit (4 weeks).
  Assessed using the Mini-mental state examination at baseline, discharge and follow-up visit. If the participant is not discharged after 4 weeks the follow-up will be examined at the hospital.
Strength, Assistance in walking, Rise from a chair, Climb stairs, and Falls (SARC-F) questionnaire. | Baseline to follow-up visit (4 weeks).
  Assessed at baseline, discharge and follow-up visit using the questionnaire Strength, Assistance in walking, Rise from a chair, Climb stairs, and Falls (SARC-F).
Perceived health - Health-related Quality of Life questionnaire (Euroqol EQ-5D-5L) | Baseline to follow-up visit (4 weeks).
  Assessed at baseline, discharge and follow-up visit using the questionnaire Health-related Quality of Life questionnaire (Euroqol EQ-5D-5L).
Perceived health - Brief Illness Perception Questionnaire (BIPQ) | Baseline to follow-up visit (4 weeks).
  Assessed at baseline, discharge and follow-up visit using the questionnaire Brief Illness Perception Questionnaire (BIPQ).
Dual Energy X-Ray Absorptiometry - Appendicular lean mass | Follow-up visit (4 weeks).
  Difference between exercise and control group in appendicular lean mass assessed at the 4-week follow-up using dual energy x-ray absorptiometry.
Dual Energy X-Ray Absorptiometry - Percentage of body fat | Follow-up visit (4 weeks).
  Difference between exercise and control group in percentage of body fat assessed at the 4-week follow-up using dual energy x-ray absorptiometry.
Dual Energy X-Ray Absorptiometry - Android fat | Follow-up visit (4 weeks).
  Difference between exercise and control group in android fat assessed at the 4-week follow-up using dual energy x-ray absorptiometry.
Dual Energy X-Ray Absorptiometry- Gynoid fat | Follow-up visit (4 weeks).
  Difference between exercise and control group in gynoid fat assessed at the 4-week follow-up using dual energy x-ray absorptiometry.
Rectus femoris cross-sectional area | Baseline to follow-up visit (4 weeks).
  Change in cross-sectional area assessed at baseline, discharge and 4-week follow-up using an ultrasound of rectus femoris in the dominant leg. If the participant is not discharged after 4 weeks, only baseline and follow-up will be assessed. It will be measured at the distal third and midpoint between the anterior superior iliac spine and the proximal point of the patella.
Rectus femoris echo intensity | Baseline to follow-up visit (4 weeks).
  Change in echo intensity of rectus femoris assessed at baseline, discharge and 4-week follow-up using skeletal muscle ultrasound in the dominant leg. If the participant is not discharged after 4 weeks, only baseline and follow-up will be assessed. It will be measured at the distal third and midpoint between the anterior superior iliac spine and the proximal point of the patella.
Rectus femoris echo variation | Baseline to follow-up visit (4 weeks).
  Change in echo variation of rectus femoris assessed at baseline, discharge and 4-week follow-up using skeletal muscle ultrasound in the dominant leg. If the participant is not discharged after 4 weeks, only baseline and follow-up will be assessed. It will be measured at the distal third and midpoint between the anterior superior iliac spine and the proximal point of the patella.
Rectus femoris pennation angle | Baseline to follow-up visit (4 weeks).
  Change in pennation angle of rectus femoris assessed at baseline, discharge and 4-week follow-up using skeletal muscle ultrasound in the dominant leg. If the participant is not discharged after 4 weeks, only baseline and follow-up will be assessed. It will be measured at the distal third and midpoint between the anterior superior iliac spine and the proximal point of the patella.
Thickness of the anterior thigh muscles | Baseline to follow-up visit (4 weeks).
  Change in anterior thigh muscle thickness assessed at baseline, discharge and 4-week follow-up, measured from the mid-anterior point rectus femoris to the mid posterior point of vastus intermedius of the femoral quadriceps in the dominant leg. If the participant is not discharged after 4 weeks, only baseline and follow-up will be assessed. It will be measured at the distal third and midpoint between the anterior superior iliac spine and the proximal point of the patella.
Thickness of rectus femoris | Baseline to follow-up visit (4 weeks).
  Change in rectus femoris muscle thickness assessed at baseline, discharge and 4-week follow-up, measured from the mid-anterior point rectus femoris to the mid posterior point in the dominant leg. If the participant is not discharged after 4 weeks, only baseline and follow-up will be assessed. It will be measured at the distal third and midpoint between the anterior superior iliac spine and the proximal point of the patella.
Bioelectrical Impedance - Appendicular lean body mass | Baseline to follow-up visit (4 weeks).
  Change in estimated appendicular lean body mass using bioelectrical impedance assessed at baseline, discharge and 4-week follow-up. If the participant is not discharged after 4 weeks, only baseline and follow-up will be assessed.
Bioelectrical Impedance - Total lean body mass | Baseline to follow-up visit (4 weeks).
  Change in estimated total lean body mass using bioelectrical impedance assessed at baseline, discharge and 4-week follow-up. If the participant is not discharged after 4 weeks, only baseline and follow-up will be assessed.
Bioelectrical Impedance - Percentage of body fat | Baseline to follow-up visit (4 weeks).
  Change in estimated percentage of body fat using bioelectrical impedance assessed at baseline, discharge and 4-week follow-up. If the participant is not discharged after 4 weeks, only baseline and follow-up will be assessed.
Readmission rates. | Baseline until 1 year follow-up.
  Time-to-event, number of events and number of days and reason for event will be assessed. The event will be assessed at 30 days post-discharge, 90 days post-discharge, and 1 year post intervention.
Sick leave rates. | Baseline until 1 year follow-up.
  Time-to-event, number of events and number of days and reason for event will be assessed. The event will be assessed at 30 days post-discharge, 90 days post-discharge, and 1 year post intervention
All cause mortality | Baseline until 1 year follow-up.
  Time-to-event, number of events and number of days and reason for event will be assessed. The event will be assessed during hospitalization, 30 days post-discharge, 90 days post-discharge, and 1 year post intervention.
Use of antidiabetic medication 1-year post inclusion | Baseline until 1 year follow-up.
  The use of which types of antidiabetic medication will be assessed at baseline, discharge, and 1-year follow up.
Circulatory factors in plasma - Interferon-γ | Baseline to follow-up visit (4 weeks).
  Change in plasma Interferon-γ assessed using the Meso Scale Discovery's V-PLEX Proinflammatory Panel 1 Human Kit. These samples will be conducted at baseline, discharge, and follow-up visit. If the participant is not discharged within 4 weeks, samples will only be collected at baseline and follow-up.
Circulatory factors in plasma - Interleukin-1β | Baseline to follow-up visit (4 weeks).
  Change in plasma interleukin-1β assessed using the Meso Scale Discovery's V-PLEX Proinflammatory Panel 1 Human Kit. These samples will be conducted at baseline, discharge, and follow-up visit. If the participant is not discharged within 4 weeks, samples will only be collected at baseline and follow-up.
Circulatory factors in plasma - Interleukin-2 | Baseline to follow-up visit (4 weeks).
  Change in plasma interleukin-2 assessed using the Meso Scale Discovery's V-PLEX Proinflammatory Panel 1 Human Kit. These samples will be conducted at baseline, discharge, and follow-up visit. If the participant is not discharged within 4 weeks, samples will only be collected at baseline and follow-up.
Circulatory factors in plasma - Interleukin-4 | Baseline to follow-up visit (4 weeks).
  Change in plasma interleukin-4 assessed using the Meso Scale Discovery's V-PLEX Proinflammatory Panel 1 Human Kit. These samples will be conducted at baseline, discharge, and follow-up visit. If the participant is not discharged within 4 weeks, samples will only be collected at baseline and follow-up.
Circulatory factors in plasma - Interleukin-6 | Baseline to follow-up visit (4 weeks).
  Change in plasma interleukin-6 assessed using the Meso Scale Discovery's V-PLEX Proinflammatory Panel 1 Human Kit. These samples will be conducted at baseline, discharge, and follow-up visit. If the participant is not discharged within 4 weeks, samples will only be collected at baseline and follow-up.
Circulatory factors in plasma - Interleukin-8 | Baseline to follow-up visit (4 weeks).
  Change in plasma interleukin-8 assessed using the Meso Scale Discovery's V-PLEX Proinflammatory Panel 1 Human Kit. These samples will be conducted at baseline, discharge, and follow-up visit. If the participant is not discharged within 4 weeks, samples will only be collected at baseline and follow-up.
Circulatory factors in plasma - Interleukin-10 | Baseline to follow-up visit (4 weeks).
  Change in plasma interleukin-8 assessed using the Meso Scale Discovery's V-PLEX Proinflammatory Panel 1 Human Kit. These samples will be conducted at baseline, discharge, and follow-up visit. If the participant is not discharged within 4 weeks, samples will only be collected at baseline and follow-up.
Circulatory factors in plasma - Interleukin-12p70 | Baseline to follow-up visit (4 weeks).
  Change in plasma interleukin-12p70 assessed using the Meso Scale Discovery's V-PLEX Proinflammatory Panel 1 Human Kit. These samples will be conducted at baseline, discharge, and follow-up visit. If the participant is not discharged within 4 weeks, samples will only be collected at baseline and follow-up.
Circulatory factors in plasma - Interleukin-13 | Baseline to follow-up visit (4 weeks).
  Change in plasma interleukin-13 assessed using the Meso Scale Discovery's V-PLEX Proinflammatory Panel 1 Human Kit. These samples will be conducted at baseline, discharge, and follow-up visit. If the participant is not discharged within 4 weeks, samples will only be collected at baseline and follow-up.
Circulatory factors in plasma - Tumor Necrosis Factor-α | Baseline to follow-up visit (4 weeks).
  Change in plasma tumor necrosis factor-α assessed using the Meso Scale Discovery's V-PLEX Proinflammatory Panel 1 Human Kit. These samples will be conducted at baseline, discharge, and follow-up visit. If the participant is not discharged within 4 weeks, samples will only be collected at baseline and follow-up.
Circulatory factors in plasma - Myostatin | Baseline to follow-up visit (4 weeks).
  Change in plasma myostatin assessed using a Meso Scale custom plate. These samples will be conducted at baseline, discharge, and follow-up visit. If the participant is not discharged within 4 weeks, samples will only be collected at baseline and follow-up.
Circulatory factors in plasma - Follistatin | Baseline to follow-up visit (4 weeks).
  Change in plasma follistatin assessed using a Meso Scale custom plate. These samples will be conducted at baseline, discharge, and follow-up visit. If the participant is not discharged within 4 weeks, samples will only be collected at baseline and follow-up.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Copenhagen University Hospital, Copenhagen, Capitol Region of Denmark
  - Departement of Infectious Diseases - Hvidovre Hospital, Copenhagen, Capitol Region of Denmark

IPD SHARING:
Plan to Share IPD: No
If the data can be fully anonymized the researchers will consider to share the data